CLINICAL TRIAL: NCT02542891
Title: E-Compared: Comparative Effectiveness Research on Internet Based Depression Treatment- French Trial
Brief Title: European Comparative Effectiveness Research on Internet-based Depression Treatment
Acronym: E-COMPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Commission (Other); Fondation FondaMental (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C15-16
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2016-12

CONDITIONS: Depressive Disorder
Keywords: e-health; depressive disorder; cost-effectiveness; Cognitive behavioral treatment
MeSH Terms: conditions — Depressive Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blended CBT (Experimental): Internet based blended depression treatment combines individual face-to-face cognitive behavioural therapy (CBT) with CBT delivered through an Internet based treatment platform with smart phone components. The core components of the CBT treatment are: (1) psycho-education, (2) cognitive restructuring, (3) behavioural activation, and (4) relapse prevention. These will be delivered over 16 sessions (8 online and 8 face-to-face), once a week. The online platform is called Moodbuster.
  The trial will not interfere with regular medication treatment, and patient's care will be monitored throughout the study.
  Interventions: Other: Blended CBT
- Treament as Usual (TAU) (Active Comparator): In order to increase the comparability between the two arms, we defined TAU as a traditional face to face CBT of 16 sessions. These sessions will be administered over a course of 16 weeks.
  The trial will not interfere with regular medication treatment, and patient's care will be monitored throughout the study.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: Blended CBT
  Other Names: Moodbuster Platform
  Arms: Blended CBT
Other: Treatment as Usual (TAU)
  Arms: Treament as Usual (TAU)

SUMMARY:
To compare the clinical impact and cost-effectiveness of blended Cognitive Behavioural Therapy (CBT) for adults with major depressive disorder (MDD) with treatment as usual (TAU). Within the French context the TAU is considered as the traditional face to face CBT.

DETAILED DESCRIPTION:
Background:

Depression is a common mental disorder with a negative impact on mental well-being, quality of life, and social and work-related functioning both in the short and longer term. Additionally, depression is associated with increased morbidity, mortality, health care utilization and health care costs. On a population level, depression is one of the most costly diseases. The economic costs of depression were estimated at €136.3 billion (EU25) in 2010 in the EU and are still rising. European health care systems face the challenge of improving access to cost-effective treatments while simultaneously working to sustain budgetary stability in times of economic austerity.

Internet-based depression treatment appears a very promising alternative to current routine depression treatment strategies. Meta-analyses have demonstrated the clinical effectiveness and potential cost-effectiveness of Internet-based treatment for depression in controlled research setting. Internet-based treatment thus has the potential to keep depression treatment affordable, as it enables mental health care providers to reach out to large populations needing depression treatment at a better cost-effectiveness than those of standard treatment as usual (TAU), but with similar levels of clinical efficacy and quality of care. The trials will be conducted in 8 European countries.

Objective:

To compare the clinical impact and cost-effectiveness of blended Cognitive Behavioural Therapy (CBT) for adults with major depressive disorder (MDD) with treatments as usual (TAU)-face to face CBT in expert centres specialized in depression.

Study design:

The study is a two-arm randomized controlled non-inferiority and cost-effectiveness trial. The trial will be conducted in expert centres in France. A total of 150 patients with MDD will be assigned to one of two treatment arms: 1) blended CBT, 2) TAU. Respondents in both arms will be followed until 12 months after baseline (measures will be taken at baseline, 3 months, post- treatment (17 weeks), 6 months and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Meet DSM-IV diagnostic criteria for MDD confirmed by MINI International Neuropsychiatric Interview version 5.0
* Having a PHQ-9 score greater than 5
* Having access to a PC and Internet connection
* Having ( or accepting to be loaned) a smartphone that is compatible with the mobile component of the intervention
* Understanding of the French language spoken and written

Exclusion Criteria:

* Current high risk for suicide according to the MINI Interview section C
* Serious psychiatric co-morbidity: substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, and suicide risks, as established at the MINI interview
* Currently receiving psychological treatment for depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10-31 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 12 months
  The primary outcome measure is symptoms of depression as assessed with Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001). The PHQ-9 is a nine-item mood module that can be used to screen and to diagnose patients with depressive disorders. The 9 items are each scored on a 0-3 scale with the total score ranging from 0-27 and higher scores indicating more severe depression. The PHQ-9 has shown to have good psychometric properties (Wittkampf, Naeije, Schene, Huyser, & van Weert, 2007).

SECONDARY OUTCOMES:
QIDS-SR16 | 12 months
  The 16 item self-report version of the Quick Inventory of Depressive Symptomatology Self-Report (QIDS-16-SR) US Translation (Rush et al., 2003) is used in addition to the PHQ-9 because it is a promising questionnaire for assessing depressive symptoms especially in specialized mental health care whereas the PHQ-9 is developed for use in primary care.The QIDS is a questionnaire that screens for depressive symptoms and assesses depression severity. The QIDS is available in both clinician-rated (IDS-C) and patient self-report (IDS-SR) forms. The QIDS consists of 16 items (each item scores 0-3) and includes symptom domains of MDD based on DSM-IV and Research Diagnostic Criteria (RDC).
M.I.N.I | 12 months
  The full M.I.N.I. 5.0,with exception of section M (Anorexia Nervosa), N (Bulimia nervosa), and P (Antisocial personality disorder), will be assessed at baseline to assess lifetime and current depression, and current comorbid disorders that often co-occur with and predict the onset of depression (anxiety disorders and PTSD) and other comorbid disorders that are an exclusion criteria in this study (i.e. substance dependence, bipolar affective disorder, psychotic illness, and obsessive compulsive disorder). At 12 months follow-up, the depression, anxiety and PTSD sections will be assessed again.
MADRS | 12 months
  The MADRS (Montgomery and Asberg Depression Rating Scale) is a hetero-assessment of depressive symptoms evaluated by clinicians.

OTHER OUTCOMES:
EQ-5D-5L | 12 months
  Quality of life will be assessed with the EQ-5D-5L (EuroQol).The EQ-5D-5L is a self-report questionnaire which measures health related quality of life and enables conversion to utility scores to calculate Quality-Adjusted Life-Years (QALYs). The EQ-5D-5L consists of five dimensions: mobility, self-care, ordinary activities, discomfort, and mood state related to anxiety or depression. Each item consists of five categories ranging from no problems to a lot of problems (Van Agt, Essink-Bot, Krabbe, & Bonsel, 1994).
AQOL-6D | 12 months
  Health-Related Quality of Life will optionally be measured with the Assessment of Quality of Life instrument (AQoL) (Hawthorne, Richardson, & Osborne, 1999). For the current study the AQoL-6D (Richardson, Peacock, Hawthorne, Lezzi, Elsworth, & Day, 2012) which consists of 20 questions measured on a 5 point scale will be used. The AQoL-6D includes the six dimensions: independent living, mental health, coping, relationships, pain, and senses.
TIC-P | 12 months
  Health service uptake and production loss due to illness will be measured with the Trimbos and iMTA Questionnaires on Costs Associated with Psychiatric Illness (TiC-P; Hakkaart-van Rooijen, van Straten, Donker, Tiemens, 2002). The TiC-P is a self-report questionnaire and consists of two different parts that can be administrated separately. Part I will be used to assess the participants' healthcare utilization and medication use. Part II (short form health and labor questionnaire [SF-HLQ]) measures lost productivity costs resulting from absenteeism (being absent from work because of illness) and presenteeism (being present at work while ill which may lead to reduced efficiency) and consists of 11 items. Healthcare utilization and productivity losses will be valued using country-specific prices.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Chevreul, Dr, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (10):
- France (10):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - CHU de Brest, Brest
  - Centre Hospitalier Le Vinatier-, Bron
  - CHU de Clermont- Ferrnand, Clermont-Ferrand
  - Hôpital A. Chenevier, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital de la conception Pôle Psychiatrie Centre, Marseille
  - CHRU Lapeyronie, Montpellier
  - Hôptial Fernand Widal, Paris
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] van Genugten CR, Schuurmans J, Hoogendoorn AW, Araya R, Andersson G, Banos R, Botella C, Cerga Pashoja A, Cieslak R, Ebert DD, Garcia-Palacios A, Hazo JB, Herrero R, Holtzmann J, Kemmeren L, Kleiboer A, Krieger T, Smoktunowicz E, Titzler I, Topooco N, Urech A, Smit JH, Riper H. Examining the Theoretical Framework of Behavioral Activation for Major Depressive Disorder: Smartphone-Based Ecological Momentary Assessment Study. JMIR Ment Health. 2021 Dec 6;8(12):e32007. doi: 10.2196/32007. PMID 34874888
- [Derived] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181